CLINICAL TRIAL: NCT06455761
Title: 68Ga-DOTA-NI-FAPI04 PET/CT in Patients With Various Types of Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FirstAHFujian-68Ga-FAPI
Record Dates: First submitted 2024-06-07; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 68Ga-DOTA-NI-FAPI04 PET/ CT (Experimental): Intravenous injection of one dosage of 111-148 MBq (3-4 mCi) 68Ga-DOTA-NI-FAPI04. Tracer doses of 68Ga-DOTA-NI-FAPI04 will be used to detect tumors by PET/CT.
  Interventions: Drug: 68Ga-DOTA-NI-FAPI04
- 68Ga-FAPI/18F-FDG PET/ CT (Experimental): Intravenous injection of one dosage of 111-148 MBq (3-4 mCi) 68Ga-FAPI or 3.7 MBq (0.1 mCi)/Kg 18FFDG. Tracer doses of 68Ga-FAPI/18F-FDG will be used to detect tumors by PET/CT.
  Interventions: Drug: 68Ga-FAPI/18F-FDG

INTERVENTIONS:
Drug: 68Ga-DOTA-NI-FAPI04 — Intravenous injection of one dosage of 111-148 MBq (3-4 mCi) 68Ga-DOTA-NI-FAPI04. Tracer doses of 68Ga-DOTA-NI-FAPI04 will be used to detect tumors by PET/CT.
  Arms: 68Ga-DOTA-NI-FAPI04 PET/ CT
Drug: 68Ga-FAPI/18F-FDG — Intravenous injection of one dosage of 111-148 MBq (3-4 mCi) 68Ga-FAPI or 3.7 MBq (0.1 mCi)/Kg 18F-FDG. Tracer doses of 68Ga-FAPI/18F-FDG will be used to detect tumors by PET/CT.
  Arms: 68Ga-FAPI/18F-FDG PET/ CT

SUMMARY:
As a novel radiotracer targeting fibroblast activation protein (FAP), 68Ga-DOTA-NI-FAPI04 is a novel agent incorporating a hypoxia sensitive nitroimidazole(NI)-moiety and a FAP-targeting. In this study, we observed the diagnostic performance of 68Ga-DOTA-NI-FAPI04 PET/CT in patients with different types of cancer, and compared its imaging results with those of 68Ga-FAPI or 18F-FDG PET/CT.

DETAILED DESCRIPTION:
Carcinoma-associated fibroblasts (CAFs) are an integral part of the tumor microenvironment, and fibroblast activation protein (FAP), as a specific marker of CAFs, is overexpressed in more than 90% of epithelial malignant tumors' CAFs, with limited expression in normal tissues, making it an appropriate target for various tumors. Currently, several tracers targeting FAP for diagnostic purposes have been developed, such as 68Ga-FAPI-04, 68Ga-FAPI-02, showing high efficacy in tumor staging and restaging. As a novel radiotracer targeting fibroblast activation protein (FAP), 68Ga-DOTA-NI-FAPI04 is a novel agent incorporating a hypoxia sensitive nitroimidazole(NI)-moiety and a FAP-targeting. In this study, we observed the diagnostic performance of 68Ga-DOTA-NI-FAPI04 PET/CT in patients with different types of cancer, and compared its imaging results with those of 68Ga-FAPI or 18F-FDG PET/CT.

ELIGIBILITY:
Inclusion Criteria:

Various solid tumors with available histopathological findings; Signed informed consent.

Exclusion Criteria:

pregnant or lactational women; who suffered from severe hepatic and renal insufficiency.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value | through study completion, an average of 3 months
  Sensitivity and Specificity of 68Ga-DOTA-NI-FAPI04 in Patients With Various Types of Cancer and comrare it with 68Ga-FAPI/18F-FDG PET/CT.

SECONDARY OUTCOMES:
SUV of tumors | through study completion, an average of 3 months
  Compare the SUV of tumors between 68Ga-DOTA-NI-FAPI04 PET/CT and 68Ga-FAPI/18F-FDG PET/CT.

CONTACTS AND LOCATIONS:
Overall Officials: Weibing Weibing, MD, Principal Investigator — First Affiliated Hospital of Fujian Medical University
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, China